CLINICAL TRIAL: NCT01795898
Title: Efficacy, Safety and Quality of Life Outcome of Fentanyl Transdermal Patch (Durogesic-D-Trans) Among Filipino Patients With Osteoarthritis and Chronic Low Back Pain
Brief Title: An Efficacy and Safety Study of Fentanyl Transdermal Patch in Filipino Participants With Osteoarthritis and Chronic Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015268; FENPAI4074
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Results first posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-06

CONDITIONS: Osteoarthritis; Low Back Pain
Keywords: Osteoarthritis; Low back pain; Fentanyl transdermal patch; Durogesic-D-Trans
MeSH Terms: conditions — Osteoarthritis; Low Back Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fentanyl transdermal patch (Experimental): Fentanyl transdermal patches releasing 12.5 microgram of fentanyl will be applied for 3 days. The patches will be replaced every 3 days (Day 3, 7 and 10).
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Fentanyl transdermal patches releasing 12.5 microgram of fentanyl will be applied for 3 days. The patches will be replaced every 3 days (Day 3, 7 and 10).
  Other Names: DUROGESIC-D-TRANS

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of fentanyl among Filipino participants with osteoarthritis (disorder which is seen mostly in older persons in which the joints become painful and stiff) and chronic (lasting a long time) low back pain.

DETAILED DESCRIPTION:
This is an open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving, "unblinded") single-arm and prospective study (study following participants forward in time) of fentanyl in participants with osteoarthritis and Chronic low back pain with moderate (medium level of seriousness) and severe (very serious, life threatening) pain levels. Participants will be treated with fentanyl transdermal patch (patch containing a drug that is put on the skin so the drug will enter the body through the skin) starting with 12.5 microgram (mcg) dose of fentanyl. The dose will be increased on Day 3, if needed, by 12.5 mcg. Dose adjustments will be done every 3 days. Maximum of 50 mcg dose of fentanyl will be allowed. Participants will be evaluated for pain levels and quality of life using Brief pain inventory (BPI) score and Clinical global impression-severity (CGI-S) score. Tramadol 50 milligram tablet at a maximum of 6 tablets per day will be used as supplemental doses of analgesic (drug used to control pain). Participants' safety will be monitored through out the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with osteoarthritis and chronic low back pain
* 3 months of persistent moderate to severe pain levels
* More than 3 times a week frequency or daily moderate to severe pain
* Moderate to severe pain at Baseline (at least a score of 4 in the 11-point numerical pain scale) Exclusion Criteria
* History of allergy to fentanyl transdermal patch or its components and history of illicit drug use for the past 3 months
* Active skin disease preventing application of the transdermal system
* Chronic pulmonary disease (lung disorder)
* Participants susceptible to intracranial (inside the skull) effects of carbon dioxide retention
* Pregnant and breastfeeding mothers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical trial, Study Director — Janssen Pharmaceutica
Locations (1):
- Quezon City, Philippines

RESULTS

PARTICIPANT FLOW:
Groups:
- Fentanyl: Fentanyl transdermal (through the skin) patches releasing 12.5 microgram (mcg) of fentanyl were applied for 3 days. The patches were replaced every 3 days (Day 3, 7 and 10) with an increase in dose by 12.5 mcg to a maximum of 50 mcg.
Period: Overall Study
Arm/Group | Fentanyl
Started | 237
Completed | 177
Not Completed | 60
Not completed — Adverse Event | 27
Not completed — Lost to Follow-up | 20
Not completed — Withdrawal of consent | 6
Not completed — Diagnosed with metastasis | 1
Not completed — No pain | 1
Not completed — Death | 1
Not completed — Withdrew consent & had adverse events | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Fentanyl: Fentanyl transdermal patches releasing 12.5 mcg of fentanyl were applied for 3 days. The patches were replaced every 3 days (Day 3, 7 and 10) with an increase in dose by 12.5 mcg to a maximum of 50 mcg.
Arm/Group | Fentanyl
Number analyzed (Participants) | 237
Age Continuous [Mean (Standard Deviation); unit: Years] | 48.202 (11.137)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174
  Male | 63
Number of Participants With Clinical Global Impression-Improvement (CGI-I) Score: Clinician [Number; unit: Participants] — CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. Here, 'N' signifies the participants analyzed for this study specific Baseline characteristic and is Intent-to-treat population defined as all the participants who received at least 1 dose of study medication and had at least 1 follow-up visit with assessment=203.
  Participants
    Not evaluated | 46
    No change | 21
    Minimally improved | 38
    Much improved | 93
    Very Much improved | 5
Number of Participants With Clinical Global Impression-Improvement (CGI-I) Score: Participant [Number; unit: Participant] — CGI-I is a 7-point scale that requires the participant to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. Number of participants analysed for this study specific Baseline characteristic=203.
  Participant
    Not evaluated | 46
    No change | 21
    Minimally improved | 40
    Much improved | 88
    Very Much improved | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Severity Score at Day 30
Description: BPI is an 11-item self-report questionnaire that is designed to assess the severity and impact of pain on daily functions. BPI- severity consists of 4 questions (items) that assess pain intensity (worst, least, average, right now). Each question (item) is answered on a scale ranging from 0 to 10; '0=No pain and 10=Pain as bad as you can imagine'. Measure can be scored by item, with lower scores being indicative of less pain or pain interference. Change: Score at Day 30 minus score at Baseline.
Time Frame: Baseline and Day 30
Population: The intent-to-treat (ITT) population was defined as all the participants who received at least 1 dose of study medication and had at least 1 follow-up visit with assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl
Number analyzed (Participants) | 203
Units on a scale
  Baseline: Worst | 7.20 (1.922)
  Baseline: Least | 3.83 (1.904)
  Baseline: Average | 5.59 (1.682)
  Baseline: Right now | 5.49 (2.121)
  Change at Day 30: Worst | -5.000 (2.661)
  Change at Day 30: Least | -3.049 (2.124)
  Change at Day 30: Average | -4.246 (2.096)
  Change at Day 30: Right now | -4.404 (2.464)

2. Primary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Interference Score at Day 30
Description: BPI is an 11-item self-report questionnaire that is designed to assess the severity and impact of pain on daily functions. BPI-interference consists of 7 questions (items) that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each question (item) is answered on a scale ranging from 0 to 10; '0=No pain and 10=Pain as bad as you can imagine'. Measure can be scored by item, with lower scores being indicative of less pain or pain interference. Change: Score at Day 30 minus score at Baseline.
Time Frame: Baseline and Day 30
Population: The ITT population was defined as all the participants who received at least 1 dose of study medication and had at least 1 follow-up visit with assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl
Number analyzed (Participants) | 203
Units on a scale
  Baseline: General activity | 5.73 (2.020)
  Baseline: Mood | 4.94 (2.288)
  Baseline: Walking ability | 5.25 (2.417)
  Baseline: Normal work | 5.34 (2.242)
  Baseline: Relationship w/others | 4.33 (2.345)
  Baseline: Sleep | 5.05 (2.430)
  Baseline: Enjoyment of life | 4.71 (2.513)
  Change at Day 30: General activity | -4.502 (2.470)
  Change at Day 30: Mood | -4.118 (2.487)
  Change at Day 30: Walking ability | -4.182 (2.618)
  Change at Day 30: Normal work | -4.251 (2.504)
  Change at Day 30: Relationship w/others | -3.700 (2.486)
  Change at Day 30: Sleep | -4.355 (2.639)
  Change at Day 30: Enjoyment of life | -3.966 (2.611)

3. Primary Outcome: Number of Participants Requiring Rescue Medication
Description: Rescue medications are periodic supplemental doses of analgesic which might be required to control pain. Tramadol 50mg tablet at a maximum of 6 tablets per day was used as standard rescue medication.
Time Frame: Day 30
Population: All participants suffering from osteoarthritis (disorder, which is seen mostly in older persons, in which the joints become painful and stuff) and chronic (lasting a long time) low back pain and who took at least 1 dose of study medication and had at least 1 follow-up visit during the study.
Measure: Number; unit: Participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 237
Participants | 41

4. Primary Outcome: Number of Participants With Clinical Global Impression-Improvement (CGI-I) Score: Clinician
Description: CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: Day 30
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 203
Participants
  Very much worse | 1
  No change | 5
  Minimally improved | 16
  Much improved | 30
  Very Much improved | 151

5. Primary Outcome: Number of Participants With Clinical Global Impression-Improvement (CGI-I) Score: Participant
Description: CGI-I is a 7-point scale that requires the Participant to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: Day 30
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 203
Participants
  Very much worse | 1
  Minimally worse | 1
  No change | 5
  Minimally improved | 14
  Much improved | 33
  Very Much improved | 149

ADVERSE EVENTS:
Time Frame: Baseline up to Day 30
Arm/Group | Fentanyl
Serious Adverse Events (participants affected / at risk) | 5/237
Other Adverse Events (participants affected / at risk) | 156/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Fentanyl (N=237)
Nausea (Gastrointestinal disorders) | 2
Aneurysm ruptured (Vascular disorders) | 1/1
Vomiting (Gastrointestinal disorders) | 2
Bradycardia (Cardiac disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl (N=237)
Dizziness (General disorders) | 128
Nausea (General disorders) | 92
Vomiting (General disorders) | 61
Somnolence (General disorders) | 39
Pruritus (General disorders) | 13
Insomnia (General disorders) | 5
Headache (General disorders) | 4
Palpitation (General disorders) | 3
Rashes (General disorders) | 3
Weakness (General disorders) | 3
Chest pain (General disorders) | 2
Cold clammy perspiration (General disorders) | 2
Flushing (General disorders) | 2
Muscle trembling (General disorders) | 2
Arm heaviness (General disorders) | 1
Blurring of vision (General disorders) | 1
Chills (General disorders) | 1
Constipation (General disorders) | 3
Dryness of mouth (General disorders) | 1
Dyspepsia (General disorders) | 1
Hematoma (General disorders) | 1
Hypertension (General disorders) | 1
Swelling of both ankles (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No